CLINICAL TRIAL: NCT07064044
Title: Effects of Muscle Energy Technique With and Without Patellar Inferior Glide on Pain, Range of Motion and Disability in Patients With Patellofemoral Pain Syndrome
Brief Title: Muscle Energy Technique With and Without Patellar Inferior Glide in Patients With Patellofemoral Pain Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/24/0162 Tayba
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Pain; Disability; Range of motion
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle Energy Technique and Patellar Inferior Glide (Experimental): Muscle Energy Technique for Hamstrings and Quadriceps While the patient contract muscle (Hamstring / Quadriceps) the therapist applies a gentle controlled force. After the contraction patient release and the therapist reposition the leg into a new barrier. Intensity of contraction will be 20-25-% of maximum strength. Each contraction will be held for 5-7 seconds, followed by additional passive stretching maintained for 30 and the relaxation patellar inferior glide applied at patella: the examiner applied a gentle downward force on the patella with their right hand, while the left hand controlled the direction of the patella's movement. This will be applied for 3-4 minutes as tolerated by the patient.
  Interventions: Other: Muscle Energy Technique and Patellar Inferior Glide
- Conventional Physiotherapy treatment (Active Comparator): TENS applied, Ultrasound therapeutic modality applied, Hip and knee muscles strengthening exercises
  Interventions: Other: Conventional Traetment

INTERVENTIONS:
Other: Conventional Traetment — TENS applied for 10 minutes, Therapeutic ultrasound,Hip abductors and lateral rotators strengthening, Hamstring muscle passive stretching, Isometrics for quadriceps, given thrice a week for 4 weeks .
  Arms: Conventional Physiotherapy treatment
Other: Muscle Energy Technique and Patellar Inferior Glide — Muscle Energy Technique for Hamstrings and Quadriceps While the patient contract muscle (Hamstring / Quadriceps) the therapist applies a gentle controlled force. After the contraction patient release and the therapist reposition the leg into a new barrier. Intensity of contraction will be 20-25-% of maximum strength. Each contraction will be held for 5-7 seconds, followed by additional passive stretching maintained for 30 and the relaxation patellar inferior glide applied at patella: the examiner applied a gentle downward force on the patella with their right hand, while the left hand controlled the direction of the patella's movement. This will be applied for 3-4 minutes as tolerated by the patient.
  Arms: Muscle Energy Technique and Patellar Inferior Glide

SUMMARY:
Patellofemoral pain syndrome (PFPS) is one of the most commonly diagnosed conditions among adolescents and adults with knee complaints, accounting for approximately 25% of knee disorders diagnosed in sports medical clinics. While the etiology of PFPS is suggested to be multifactorial, several contributing factors such as lower knee extensors strength, quadriceps imbalance, weak hip abductors and overuse have been identified.

DETAILED DESCRIPTION:
This study will be a randomized clinical trial and will be conducted in RIMS Rehabilitation Center Multan and Hadi Physiotherapy Center Multan. Non-probability convenient sampling will be used to collect the data. Sample size of 36 subjects with age group 20-40 years will be taken. Data will be collected from the patients having patellofemoral pain syndrome. Outcome measures will be taken using Numeric pain rating scale (NPRS) for pain, Universal Goniometer (GU) for Range of motion and Kujala Anterior Knee Pain Scale (AKPS) for disability. An informed consent will be taken. Subjects will be selected on the basis of inclusion and exclusion criteria and will be equally divided into two groups by random number generator table. Group A will receive muscle energy technique and patellar inferior glide and conventional physical therapy while group B will receive muscle energy technique and conventional treatment. Outcome measures will be measured at baseline and after 4 weeks. Data analysis will be done by SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with age 20-40Years
* Pain rating > 3 and < 7 on NPRS
* Patella alta confirmed with ISI (Insall Salvati index) ratio > 1.2 on lateral knee radiograph
* Positive Ely's test for rectus femoris tightness
* Positive eccentric step test

Exclusion Criteria:

* History of patellofemoral dislocation
* Knee osteoarthritis
* Recently undergo to surgery to knee
* Fracture in knee region
* Positive patellar tap test for knee joint effusion
* Lateral and medial tracking of patella
* Patients taking NSAIDs and corticosteroids

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | upto 4 weeks
  The Numeric Pain Rating Scale (NPRS) is perhaps the most frequently applied scale used to quantify pain intensity in the clinical setting. It is an 11-point numeric scale, ranging from 0 indicating no pain to 10 indicating worst pain imaginable
Universal Goniometer | upto 4 weeks
  Universal goniometer (UG) is commonly used as a standard method to evaluate range of motion (ROM) as part of joint motions.
Kujala Anterior Knee Pain Scale (AKPS) | upto 4 weeks
  The Kujala patellofemoral scoring system is a tool used to assess the functional ability of the knee joint, specifically in relation to patellofemoral-related issues. This scoring system ranges from 0 to 100, with higher scores indicating better knee function and less pain, while lower scores indicate greater dysfunction and more severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Samrood Akram, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Rims Rehabilitation Centre, Multan Khurd, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Widhiantari NKE, Widnyana M, Jawi IM. Risk factors of the patellofemoral pain syndrome. Kinesiology and Physiotherapy Comprehensive. 2023;2(3):74-80.
- [Background] Leon-Morillas F, Garcia-Marin M, Corujo-Hernandez C, Martin Aleman M, Castellote-Caballero Y, Cahalin LP, Infante-Guedes A, Cruz-Diaz D. Evaluating the Impact of Flossing Band Integration in Conventional Physiotherapy for Patellofemoral Pain Syndrome. J Clin Med. 2024 May 17;13(10):2958. doi: 10.3390/jcm13102958. PMID 38792499
- [Background] Abd Elhady AM, Abd Elmajeed SF, Abd Allah WA, Abd Elhamed HB. Knee Alignment-Oriented Balance Exercises Versus Conventional Balance Exercises in Treating Patellofemoral Pain Syndrome. The Egyptian Journal of Hospital Medicine (January 2024).94:975-81.
- [Background] Raju A, Jayaraman K, Nuhmani S, Sebastian S, Khan M, Alghadir AH. Effects of hip abductor with external rotator strengthening versus proprioceptive training on pain and functions in patients with patellofemoral pain syndrome: A randomized controlled trial. Medicine (Baltimore). 2024 Feb 16;103(7):e37102. doi: 10.1097/MD.0000000000037102. PMID 38363950
- [Background] Mv VK, Subramanian NB, S S, Kotamraju S, Krishnan M. Physiotherapeutic interventions on quadriceps muscle architecture in patello-femoral pain syndrome. Bioinformation. 2023 Apr 30;19(4):454-459. doi: 10.6026/97320630019454. eCollection 2023. PMID 37822824
- [Background] Veeresh G, Kumar SS, Sasidharan S. MANUAL THERAPY FOR PATELLOFEMORAL PAIN SYNDROME REVIEW OF LITERATURE. EPRA International Journal of Multidisciplinary Research (IJMR). 2024;10(5):298-309.